CLINICAL TRIAL: NCT06686004
Title: Investigating the Bioavailability of Bioactive Compounds of Vegetable (carrot) in Human Bio-fluids After Consumption
Brief Title: Bioavailability Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: Protocol Carrot-01; Not funded (Other: Newcastle University)
Record Dates: First submitted 2024-11-03; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2022-08

CONDITIONS: Absorption, Metabolism and Excretion in Healthy Volunteers; Bioavailability and AUC
Keywords: bioavailability; metabolism; carrots; carotenoids; polyacetylenes; Falcarinol; Falcarindiol; Falcarindiol-3-acetate; α-carotene; β-carotene; lutein; absorption
MeSH Terms: interventions — falcarindiol; Lutein

STUDY DESIGN:
Intervention Model Description: Active comparator: orange carrot 100g or 300g Placebo comparator: baseline - before ingestion
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose (300g) carrot with 2 slices of bread and 10g butter (Active Comparator): Test Session 2:
  The participants will consume the 300g carrots with bread and butter. This is considered a reasonable high enough dose that detection of the compounds must occur. This dose would be compared with the normal dose (100g) to see if there is more absorption of the compound when eaten a hiher dose.
  Interventions: Dietary Supplement: Carrots
- Experimental: Normal dose (100g) carrot with 2 slices of bread and 10g butter (Active Comparator): Test session 1: This is a normal dose (100g) which would be compared with the high dose to see if there dose-dependent effect in the magnitude of absorption.
  Test Session 2: All the process as in the test session 1 will be repeated for the 300g dose carrot.
  Interventions: Dietary Supplement: Carrots

INTERVENTIONS:
Dietary Supplement: Carrots — Detection of polyacetylene and carotenoids in human biofluids
  Other Names: PA: falcarinol, falcarindiol, falcarindiol-3-acetate; Carotenoids: α-carotene, β-carotene, lutein

SUMMARY:
Carrot is a unique vegetable owing to the availability of bioactive compounds polyacetylenes (PA) as well as carotenoids present in it. These compounds have been shown to be associated with reduced cancer risk in epidemiological-based studies, and also showed anticancer properties in vitro studies and in vivo in mouse and rat models. To investigate whether the PA and carotenoids could have beneficial effects in humans, the present study is designed to determine whether they are detectible in human biofluids after the ingestion of a portion of carrots and whether there is a difference in the magnitude of detection after eating a large (300g) and normal (100g) portion.

DETAILED DESCRIPTION:
The occurrence of PA and carotenoids in carrot is not a guaranteed that they have potential health benefits and biological activity in humans, as there is still insufficient knowledge as to whether they can be absorbed in human bio-fluids (blood, urine and faeces) after the food (carrot) is consumed in the literature. The bioavailability of compounds depends upon both the chemical forms and physical structures which enable a certain proportion of such compounds into circulation when introduced into the body and so are able to have an active effect.

The main goal of this trial is to investigate determine the fate of (PAs and carotenoids) found in carrots human plasma, urine and faeces.

To achieve this goal, health adult volunteers will be instructed to restrict their diet (To avoid eating food that contain the compounds of interest) for 48hrs and complete 24hr food diary.

They will fast overnight and collect urine and faecal samples on the morning of the test session. Once they arrive in the research facility, they will have fasted blood taken before eating a portion of carrots (either 100 or 300g) with bread and butter. Further blood samples will be taken at 1, 2, 4, 6, 8 and 24 hours. Urine sample will be collected at 4, 8, 12 and 24hr and up to 48hr after the carrot consumption, and faecal samples will be collected at any time the participants feel bowel movement during the study duration up to 48hr, noting the time when each sample was generated.

The participants will attend two test sessions and will be randomised to receive high (300g) and normal (100g) doses of carrot. The washout period separating the two testing sessions is at least a week.

The specific compounds of interest in this trial include PA (falcarinol, falcarindiol, and falcarindiol 3-acetate), carotenoids (α-carotene, β-carotene and lutein) and their concentrations at various time points after consumption and baseline will be measured using HPLC (for carotenoids) and LC-MS (for PA). The concentrations of the compounds at time points after ingestion will be compared with the baseline and also in relation to, normal and high carrot doses.

ELIGIBILITY:
Inclusion criteria:

* Healthy adults 20+ years old.
* Having body mass index (BMI) between ≥18.5 - ≤30 kg/m2.
* Must be willing to eat a portion (100g) of carrot in the test session 1, alongside 2 slices of bread with 10g butter.
* Must be willing to eat a portion (300g) of carrot in the test session 2, alongside 2 slices of bread with 10g butter.

Exclusion Criteria:

* Having any metabolic or gastrointestinal conditions.
* Having allergies to carrot or bread or butter.
* Taking any medication that affects metabolism or digestion.
* Smokers.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Absorption of PA and carotenoids | 48hr
  The primary outcome is testing whether a change in concentration of PA and carotenoids is seen between baseline and various time points in the biofluids after ingesting carrots.

SECONDARY OUTCOMES:
Dose-effect between the absorption of PA and carotenoids from 100g and 300g carrots | 48hr
  This is testing whether there is a difference between the high and low dose concentrations of polyacetylenes at various time points after eating carrots.

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrtition Suite, DMBB Newcastle University, Newcastle upon Tyne, Tyne and Wear, United Kingdom